CLINICAL TRIAL: NCT02617147
Title: Influence of Vitrectomy and Membrane Peeling on Choroidal Thickness
Brief Title: Choroidal Thickness Vitrectomy
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Stefan Sacu, Assoz. Prof. Priv. Doz. Dr., Medical University of Vienna
Other Study IDs: ophth04012014
Record Dates: First submitted 2015-11-24; First posted 2015-11-30 (Estimated); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Epiretinal Membrane
MeSH Terms: conditions — Epiretinal Membrane

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to assess the influence of vitrectomy on changes in central choroidea and comparing the results in imaging of the choroidea with two different OCT devices.

This is a prospective, open, non-randomized, observational, MPG study This study will be performed at the Department of Ophthalmology, Medical University of Vienna.

40 Patients who undergo vitrectomy will be included into this study. The investigation will help to gain new information about the effects of vitrectomy on the choroid.

DETAILED DESCRIPTION:
Since the development of new OCT modalities, like enhanced depth or swept-source OCT imaging, a better visualization and evaluation of retinal structures and the choroidea became possible. 23G Vitrectomy and membrane peeling seem to have an influence on posterior segment structures of the eye but data show no clear evidence evaluating those changes after surgery. Only little information is currently available on the influence or the changes resulting from vitreous surgery on the central choroidea. Hence, the aim of this study is to evaluate those influences resulting on choroidea using two different OCT devices.

To assess the influence of vitrectomy on changes in central choroidea and comparing the results in imaging of the choroidea with two different OCT devices.

This is a prospective, open, non-randomized, observational, MPG study This study will be performed at the Department of Ophthalmology, Medical University of Vienna.

40 Patients who undergo vitrectomy will be included into this study. The investigation will help to gain new information about the effects of vitrectomy on the choroid.

The measuring procedures used in this study are well tolerated and used in routine clinical practice and are non-invasive.

ELIGIBILITY:
Inclusion Criteria:

* Patients with epiretinal membrane scheduled to undergo vitrectomy without endotamponade
* Male or female, at least 18 years of age
* Written informed consent has been obtained
* Visual acuity ≥0.4

Exclusion Criteria:

* Any abnormalities preventing reliable measurements as judged by the investigator
* Participation in a clinical trial in the 3 weeks preceding the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with epiretinal membrane scheduled to undergo vitrectomy
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2014-06-16 (Actual); Primary Completion 2018-03-13 (Actual); Study Completion 2018-03-13 (Actual)

PRIMARY OUTCOMES:
choroidal thickness using 2 different OCT devices | 3 months

SECONDARY OUTCOMES:
Visual Acuity using Snellen charts | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology, Medical University of Vienna, Austria, Vienna, Austria